CLINICAL TRIAL: NCT01357473
Title: Is Hormonal Exposure of Endometrium on the First Day After Menstruation Associated With the Probability of Pregnancy in Patients Treated With Rec-FSH/ GnRH Antagonist? A Prospective Trial
Brief Title: Stop Menstruation and Pregnancy Rates in Antagonist Protocol
Status: Completed | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: DEVROEY PAUL, CRG UZ BRUSSEL
Other Study IDs: 239
Record Dates: First submitted 2011-05-09; First posted 2011-05-20 (Estimated); Last update posted 2011-05-20 (Estimated); Status verified 2011-05

CONDITIONS: Infertility
Keywords: hormonal values; menstruations; pregnancy; antagonist
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The proposal of this study is to evaluate the association between the achievement of ongoing pregnancy and hormonal levels on the first day after the period had stopped in rec-FSH/GnRH- antagonist cycles.

DETAILED DESCRIPTION:
Ovarian stimulation will be achieved by rec- FSH, Puregon® starting on day 2 of the cycle at a dose of 200 IU/day. The dose of rec-FSH remains unchanged during stimulation until day 10 of the cycle. If it is necessary to increase the dose of rec-FSH after 10 days of stimulation, or to decrease the dose of rec-FSH due to a risk of OHSS, the patient will be dropped out of the study.

To inhibit premature LH surge daily GnRH - antagonist (orgalutran 0,25mg ) is used from the morning of day 6 of stimulation.

Final oocyte maturation will be achieved by administration of 10.000 IU of HCG (Pregnyl®) as soon as ≥ 3 follicles ≥ 17 mm are present. E2 levels should not be criteria for HCG administration. Oocyte retrieval will be carried out 36 hours after HCG administration. Conventional IVF or ICSI will be carried out. Embryo transfer will be carried out day3 or day5 after oocyte retrieval.

Similar luteal support for all patients with vaginal administration of 600mg natural micronised progesterone in three separate doses (Utrogestan® 200mg 3xday) starting one day after oocyte retrieval will be used. Hormonal assessment (E2,FSH,LH,Progesterone) will be performed at initiation of stimulation, on the first day after the period had stopped and every 2 days until the day of HCG administration.

ELIGIBILITY:
Inclusion Criteria:- Age ≤ 39 years

* Body mass index between 18 and 29 kg/m²¬
* Regular cycles between 25-34 days
* Presence of both ovaries
* Basal levels of estradiol (≤ 80 pg/ml) and progesterone (≤ 1.6ng/ml) on day one of the cycle
* Treatment with IVF/ICSI
* Embryo transfer day 3 or day 5 (1 or 2 embryos)
* Patients can enter in the study only once

Exclusion Criteria:

* Presence of endometriosis stage ≥3(AFS)
* Polycystic ovarian syndrome (Rotterdam criteria)
* Need for preimplantation genetic diagnosis (PGD)
* Azoospermia testicular sperm extraction (TESE)

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Infertility women treated with rec FSH/antagonist protocol
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-02 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy rate. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: DIMITRA KYROU, MD, Principal Investigator — CRG UZ Brussel